CLINICAL TRIAL: NCT06336525
Title: Sleep Health in the Rural South and Its Relationships With Cardiometabolic Health Disparities
Brief Title: Adult Sleep Health in the Rural Appalachia and Mississippi Delta Region and Its Relationships With Cardiometabolic Health Disparities.
Status: Enrolling by invitation | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: University of Alabama at Birmingham (Other); Emory University (Other); University of Pennsylvania (Other); University of Massachusetts, Worcester (Other); The University of Texas Health Science Center at San Antonio (Other); Beth Israel Deaconess Medical Center (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Daniel J.Gottlieb, M.D.,M.P.H., Medical Doctor, Brigham and Women's Hospital
Other Study IDs: 2023P001895; R01HL164462 (NIH)
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Sleep Apnea; Insomnia; Sleep Deprivation; Sleep Disorders, Circadian Rhythm; Sleepiness, Excessive Daytime; Fatigue
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Initiation and Maintenance Disorders; Sleep Deprivation; Sleep Disorders, Circadian Rhythm; Disorders of Excessive Somnolence; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rural communities in the southern U.S. suffer a disproportionate burden of morbidity and mortality from cardiometabolic disease, with traditional risk factors explaining only a modest proportion of the excess burden of disease. There is considerable evidence that multiple dimensions of sleep health, including sleep duration, efficiency, timing, and regularity, as well as the disorders sleep apnea and insomnia, affect cardiometabolic disease risk. However, there is currently a lack of systematically developed sleep data in rural populations. The RURAL Sleep Study is an ancillary study to a recently initiated longitudinal epidemiology study in rural Appalachia and Mississippi Delta (the RURAL Study). The RURAL Sleep Study will add measures of sleep health to the complex individual, social and environmental factors and health outcome measures being evaluated by the RURAL Study, by incorporating minimally burdensome measures of multiple dimensions of sleep health. The results are expected to inform health care providers, public health officials, and the general public of the prevalence, risk factors, and consequences of impaired sleep health in these rural communities, providing a critical basis for prevention, recognition, and management of sleep disorders and improvement of sleep and cardiometabolic health.

DETAILED DESCRIPTION:
Rural communities in the southern U.S. suffer a disproportionate burden of morbidity and mortality from cardiometabolic disease, with traditional risk factors explaining only a modest proportion of the excess burden of disease. Growing evidence implicates poor sleep health as an important risk factor for cardiometabolic disease. While this is most well established for sleep apnea and insomnia, there is considerable evidence that multiple dimensions of sleep health, including sleep duration, efficiency, timing, and regularity, also affect cardiometabolic disease risk. Moreover, rural Southern communities are likely to experience high rates of impaired sleep health, reflecting high levels of psychosocial and environmental stressors, such as financial stress, social isolation, environmental pollution, and poor built environment in addition to high rates of smoking and obesity. However, there is currently a lack of systematically developed sleep data in rural populations.

Recognizing the paucity of research on cardiometabolic risk in this high-risk rural population, the NHLBI recently initiated a new longitudinal epidemiology study in rural Appalachia and Mississippi Delta (the RURAL Study) to identify the complex individual, social and environmental factors contributing to this high burden of disease. The proposed RURAL Sleep Study will complement the RURAL Study by incorporating minimally burdensome measures of multiple dimensions of sleep health at the time of baseline cohort assessment in approximately 4000 adults age 25-64 years, utilizing mobile health technologies to

1. measure sleep apnea over seven consecutive nights;
2. measure sleep duration, timing, regularity and fragmentation over multiple weeks; and
3. administer standardized questionnaires to assess insomnia, chronotype, sleep quality, sleep-related impairment, and fatigue.

These data will allow us to leverage the planned extensive assessments of cardiometabolic risk factors, subclinical disease, and psychosocial and environmental stressors (and resilience factors) to address the following specific aims:

Aim 1a. Quantify population distributions of sleep health measures in a rural cohort along dimensions of sleep apnea, insomnia, chronotype, and sleep duration, efficiency, timing, and regularity.

Aim 1b. Identify psychosocial, behavioral, and environmental correlates of sleep health in rural communities.

Aim 2. Assess the association of sleep health with cardiometabolic risk factors and subclinical cardiovascular disease independent of other established cardiovascular and metabolic risk factors.

The results are expected to inform health care providers, public health officials, and the general public of the prevalence, risk factors, and consequences of impaired sleep health in these rural communities, providing a critical basis for prevention, recognition, and management of sleep disorders and improvement of sleep and cardiometabolic health.

ELIGIBILITY:
Inclusion Criteria:

* All participants in the Risk Underlying Rural Areas Longitudinal (RURAL) Study will be eligible for enrollment in this ancillary study.

Exclusion Criteria:

* None

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will consist of a general population sample of adults age 25-64 years residing in 10 counties in the rural Appalachia and Mississippi Delta regions (AMD): Alabama, Mississippi, Louisiana, and Kentucky, with counties sampled proportional to their populations. The projected RURAL Study sample size is 4600 individuals, with approximately equal numbers in each of the four age deciles. The sample is anticipated to include 51.7% women and 48.3% men. The projected racial/ethnic make-up of the sample is 63.8% non-Hispanic white, 32.7% non-Hispanic black, 1.7% Hispanic and 1.8% other.
Sampling Method: Non-Probability Sample
Enrollment: 3680 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Oxygen desaturation index | 7 nights
  Frequency of 4% drops in nocturnal blood oxygen saturation
Insomnia Severity Index | Single measurement at baseline
  min: 0, max: 28, higher score indicates more insomnia symptoms
Sleep Duration | 3-6 months
  Mean total sleep time from accelerometry
Sleep Duration Regularity | 3-6 months
  Variability in total sleep time from accelerometry
Sleep Timing | 3-6 months
  Sleep midpoint from accelerometry
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep-related Impairment Short Form 8a | Single measurement at baseline
  raw score min: 8, max: 40; higher score indicates greater impairment

SECONDARY OUTCOMES:
Restless Legs Syndrome (RLS) | Single measurement at baseline
  Restless Legs Syndrome, yes/no
Chronotype | Single measurement at baseline
  Body's natural tendency to go to sleep and wake up at certain times
Sleep Timing Regularity | 7 days
  Variability in sleep midpoint from accelerometry
Global Sleep Quality | Single measurement at baseline
  Pittsburgh Sleep Quality Index (PSQI), min: 0, Max: 21; higher score indicates poorer sleep quality Minimum Score = 0 (better); Maximum Score = 21 (worse) Interpretation: TOTAL < 5 associated with good sleep quality TOTAL > 5 associated with poor sleep quality
Oxygen desaturation index, 3% | 7 days
  Frequency of 3% drops in nocturnal blood oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Gottlieb, MD, MPH, Principal Investigator — Brigham and Women's Hospital; Tené Lewis, PhD, Principal Investigator — Emory University; Tianyi Huang, PhD, Principal Investigator — Harvard Chan School of Public Health
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified oximetry data and the results of sleep questionnaires will be shared via the National Sleep Research Resource (NSRR) (sleepdata.org). The RURAL sleep data will be available for any researcher who provides an acceptable Data Access and Use Agreement and has appropriate regulatory approvals. The NSRR has procedures to streamline Institutional Review Board (IRB) approval (via an in house IRB process). The NSRR is in the process of migrating to Bio Data Catalyst, enabling easy linkage and interoperability with other Bio Data Catalyst data (from RURAL) and other cohorts to individuals with approved Database of Genotypes and Phenotypes (dbGaP) authorization.
  Other RURAL Study data that are integral to this project but were collected separately by the parent RURAL Study (e.g., non-sleep cardiovascular risk and outcomes data) will be distributed via RURAL Study data sharing mechanisms, including via Bio Data Catalyst and dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within one year of publication of primary study results.